CLINICAL TRIAL: NCT01661972
Title: X-TRAP: Phase I/II Study of Capecitabine Plus Aflibercept in Metastatic Colorectal Cancer
Brief Title: Phase I/II Study of Capecitabine Plus Aflibercept to Treat Metastatic Colorectal Cancer
Acronym: X-TRAP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: John Strickler, M.D. (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor-Investigator, John Strickler, M.D., Associate Professor, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Pro00037688
Record Dates: First submitted 2012-07-31; First posted 2012-08-10 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Metastatic Colorectal Cancer
Keywords: colorectal cancer; all solid tumors; metastatic; refractory; advanced solid tumors
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Capecitabine; aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1: Capecitabine and Aflibercept (Experimental): A standard 3+3 dose escalation format will be used. Capecitabine will start at 850mg/m2 to be given on days 1-14 and off days 15-21. If tolerated, the dose will then be escalated to 1000mg/m2 for the next cohort, given on the same schedule. The dose of aflibercept will be held constant at 6 mg/kg, given intravenously every 3 weeks.
  Interventions: Drug: Capecitabine and aflibercept
- Phase 2: Capecitabine and Aflibercept (Experimental): Once the RPTD of the doublet combination has been identified, an additional 50 subjects with metastatic colorectal cancer will be added to a single, Phase 2 arm
  Interventions: Drug: Capecitabine and aflibercept

INTERVENTIONS:
Drug: Capecitabine and aflibercept — Capecitabine given on days 1-14 and off days 15-21. Dose: Phase 1 cohort 1 850mg/m2 Phase 1 cohort 2 1000mg/m2, Phase 2 RPTD.
  Aflibercept will be held constant at 6 mg/kg, given intravenously every 3 weeks.
  Both agents will be administered on a 21-day cycle.

SUMMARY:
The Primary Phase I objectives are to determine the recommended phase II dose for the capecitabine and aflibercept doublet combination; and to describe any dose limiting and non-dose limiting toxicities. The Phase II Primary objective is to determine progression free survival associated with this regimen. The Phase II secondary objectives are to determine response rate associated with this regimen; to determine overall survival associated with this regimen; and to explore any correlation of clinical outcome with baseline and on treatment changes in blood-based angiogenesis biomarkers.

This open-label, non-randomized phase I/II trial is designed to assess the safety, tolerability and RPTD of capecitabine plus aflibercept in adult subjects with metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. For the phase I portion, patients must have histologically and/or cytologically confirmed malignant solid tumor that is refractory to standard therapies.

   For the phase II portion, patients must have histologically and/or cytologically confirmed metastatic colorectal carcinoma that has progressed on, is intolerant of, or is inappropriate for all standard therapies. Subjects must have been treated with a fluoropyrimidine (e.g., 5-fluorouracil or capecitabine), oxaliplatin, irinotecan and bevacizumab or have contraindication to such treatment. Prior epithelial growth factor receptor (EGFR)-targeting agent (or contraindication to these drugs) is required for subjects with K-Ras wildtype tumors
2. Measurable disease by RECIST 1.1 criteria (see Appendix 1). Previously irradiated sites can be included if there is documented progression of disease in that site.
3. Age 18 years and older.
4. KPS > 70% (see Appendix 2)
5. Life expectancy > 3 months.
6. Adequate organ and marrow function as defined below:

   * Absolute neutrophil count > 1.5 x 109/L
   * Platelet count > 100 x 109/L
   * Hemoglobin > 9 g/dl
   * Total bilirubin < 1.5 x ULN
   * AST (SGOT)/ALT (SGPT) < 2.5 x ULN (or <5 x ULN if liver metastases)
   * Creatinine clearance ≥50 mls/min by Cockcroft-Gault
   * Urine Protein/Creatinine ratio < 1 (or protein < 1+ on urinalysis or 24hour urine protein < 1gram/24 hours)
7. Previous radiotherapy for palliation of recurrent disease is allowed if >4 weeks have elapsed since completion of therapy.
8. Ability to take oral medications.
9. Ability to understand and the willingness to sign a written informed consent document.
10. Women of childbearing potential must have a negative serum pregnancy test within 7 days from day 1 of study drug; both men and women must be willing to use two methods of contraception, one of them being a barrier method during the study and for 6 months after last study drug administration.
11. Signed informed consent

Exclusion Criteria:

1. Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks from day 1 of study drug (including investigational agents, chemotherapy, radiation therapy, antibody based therapy, etc.)
2. History of severe hypersensitivity reactions/anaphylaxis attributed to humanized and/or chimeric monoclonal antibodies or other such proteins.
3. History of significant intolerance to capecitabine or 5FU (ie. Grade 4 toxicity related to one of these agents; grade 3-4 toxicity related to other concurrently administered agents is not an exclusion).
4. History of abdominal fistula or gastrointestinal perforation at any point within 6 months prior to day 1 of study drug, unless surgically repaired.
5. Active peptic ulcer disease, inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), diverticular disease or other gastrointestinal conditions with increased risk of perforation or gastrointestinal bleeding.
6. Active bleeding diathesis or history of any major bleeding, CNS bleeding, or significant hemoptysis within 6 months of enrollment.
7. Anticoagulation with warfarin (anticoagulation with low molecular weight heparin is not an exclusion).
8. History of arterial thromboembolic events or symptomatic pulmonary embolism within 6 months of study enrollment.
9. Poorly controlled hypertension [defined as systolic blood pressure (SBP of >150 mmHg or diastolic blood pressure (DBP) of >90 mmHg]
10. Patients who have had a major surgery or significant traumatic injury within 4 weeks from day 1 of study drug.
11. History of active brain metastases or carcinomatous meningitis (treated metastases are permitted, provided the patient is asymptomatic and off steroids for 28 days).
12. Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. Two acceptable forms of contraceptives must be continued throughout the trial by either sex. Hormonal contraceptives are not acceptable as a sole method of contraception. (Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to day 1 of study drug).
13. Any active infection, intercurrent illness, severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2012-08; Primary Completion 2016-06-12 (Actual); Study Completion 2016-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Strickler, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke Cancer Center, Duke University Medical Center, Durham, North Carolina
  - Virginia Oncology Associates, Norfolk, Virginia

REFERENCES:
- [Derived] Strickler JH, Rushing CN, Niedzwiecki D, McLeod A, Altomare I, Uronis HE, Hsu SD, Zafar SY, Morse MA, Chang DZ, Wells JL, Blackwell KL, Marcom PK, Arrowood C, Bolch E, Haley S, Rangwala FA, Hatch AJ, Nixon AB, Hurwitz HI. A phase Ib study of capecitabine and ziv-aflibercept followed by a phase II single-arm expansion cohort in chemotherapy refractory metastatic colorectal cancer. BMC Cancer. 2019 Nov 1;19(1):1032. doi: 10.1186/s12885-019-6234-8. PMID 31675952

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: Capecitabine is given days 1-14 of a 21 day cycle. Cohort 1 will receive 850mg/m2 Capecitabine and Cohort 2 will receive 1000mg/m2. Aflibercept 6 mg/kg is given intravenously every 3 weeks.
- Phase 2: Capecitabine at the recommended dose based on Phase 1 (850mg/m2) given on days 1-14. Aflibercept 6 mg/kg given intravenously every 3 weeks. Both agents are administered on a 21-day cycle.
Period: Overall Study
Arm/Group | Phase 1 | Phase 2
Started | 13 | 50
Completed | 11 | 46
Not Completed | 2 | 4
Not completed — Adverse Event | 1 | 2
Not completed — Death during Treatment period | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 | Phase 2 | Total
Number analyzed (Participants) | 13 | 50 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (12.3) | 57.7 (9.9) | 57.8 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 20 | 26
  Male | 7 | 30 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 14 | 16
  White | 11 | 29 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 50 | 63

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase II Dose (RPTD) for the Capecitabine and Aflibercept Doublet Combination
Description: Phase 1 of this study will be the dose escalation component to determine safety and the Recommended Phase II dose (RPTD) for the capecitabine plus aflibercept combination. Cohort 1 will receive 850mg/m2 capecitabine and 6mg/kg aflibercept. If less than 2 of 6 patients experience a dose limiting toxicity in Cohort 1, then the next patients will be enrolled in Cohort 2 at 1000mg/m2 capecitabine and 6mg/kg aflibercept. RPTD is determined by the number of dose limiting toxicities (Primary obj 2 for Phase I).
Time Frame: RPTD for the study will be determined at the completion of Phase I; up to 1 year.
Measure: Number; unit: mg/m2
Groups:
- Phase 1: Aflibercept 6 mg/kg given intravenously every 3 weeks. Capecitabine was given at 850mg/m2 for the first cohort and at 1000mg/m2 for the second cohort.
Arm/Group | Phase 1
Number analyzed (Participants) | 13
mg/m2 | 850

2. Primary Outcome: Number of Dose-Limiting Toxicities (Phase 1)
Description: Number of patients experiencing a dose-limiting toxicity in each cohort.
  A dose-limiting toxicity is defined as Grade 4 neutropenia, thrombocytopenia or anemia or grade 3 neutropenia or thrombocytopenia lasting over 7 days Grade 3 thrombocytopenia associated with bleeding Febrile Neutropenia Nausea/Vomiting or Diarrhea ≥ grade 3 and lasting ≥ 4 days despite adequate supportive measures Grade ≥ 3 Bilirubin, ALT or AST > 7 days Other non-hematologic toxicity ≥ grade 3 excluding alopecia, anorexia, fatigue, hypertension, isolated lab abnormalities (not clinically significant) and/ rare, idiosyncratic reactions to any of the study drugs. Anorexia, fatigue and hypertension will be considered as DLT only if they reach grade 4 or are considered unmanageable Treatment delay of ≥ 14 days for cycle 2 due to unresolved toxicity Treatment-related death or clinically significant,treatment-related hospitalization
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1 Cohort 1: Capecitabine 850mg/m2 given days 1-14 and off days 15-21. Aflibercept 6 mg/kg given intravenously every 3 weeks. Both agents are administered on a 21-day cycle.
- Phase 1 Cohort 2: Capecitabine 1000 mg/m2 given days 1-14 and off days 15-21. Aflibercept 6 mg/kg given intravenously every 3 weeks. Both agents are administered on a 21-day cycle.
Arm/Group | Phase 1 Cohort 1 | Phase 1 Cohort 2
Number analyzed (Participants) | 7 | 6
Participants | 1 | 2

3. Primary Outcome: Median Progression Free Survival (PFS)
Description: Time in months from the start of study treatment to the date of first progression (PD) according to the RECIST criteria, or death due to any cause. Per RECIST criteria, a PD is indicated when there is at least a 20% increase in the sum of the longest diameters from target lesions relative to the smallest sum recorded since treatment is initiated. Median PFS was estimated using a Kaplan-Meier curve, and is the time at which 50% of patients remain alive without disease progression.
Time Frame: approximately 5 months
Population: Patients enrolled in Phase 2 were included in the analysis
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Phase 2: Capecitabine at the recommended dose based on Phase 1, given days 1-14 and off days 15-21. Aflibercept 6 mg/kg given intravenously every 3 weeks. Both agents are administered on a 21-day cycle.
Arm/Group | Phase 2
Number analyzed (Participants) | 50
Months | 3.91 [2.30 to 4.47]

4. Secondary Outcome: Response Rate
Description: The percentage of patients for whom the best overall response is complete response (CR) or partial response (PR). A CR occurs when all lesions disappear; whereas, a PR is indicated when there is at least a 30% decrease in the sum of the longest diameters (LD) of the target lesion. A PD (progressive disease) occurs when there is at least a 20% increase in the sum of the LD relative to the smallest sum LD recorded since treatment is initiated. Disease is considered stable if there is no response and no PD. All patients were assigned a best response for inclusion in this calculation in accordance with the protocol.
Time Frame: approximately every 9 weeks and/or restaging, through study completion
Population: All evaluable Phase 2 patients. 5 patients were not evaluable for response and were not included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2
Number analyzed (Participants) | 45
percentage of participants | 2.22 [0.06 to 11.77]

5. Secondary Outcome: Median Survival
Description: Time in months from the start of study treatment to date of death due to any cause. Median survival was estimated using a Kaplan-Meier curve and is the time point at which 50% of patients remain alive.
Time Frame: Subjects will be followed until death which is estimated to be on average 6 months - 1 year after coming off protocol therapy
Population: Patients enrolled in Phase 2 were included in the analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2
Number analyzed (Participants) | 50
months | 7.43 [5.78 to 10.68]

ADVERSE EVENTS:
Time Frame: All serious and non-serious adverse events will be collected from time of informed consent to 30 days after a subject's last dose of study agent.
Description: Grade 2 and above adverse events for this study were collected using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Arm/Group | Phase 1 | Phase 2
Serious Adverse Events (participants affected / at risk) | 9/13 | 18/50
Other Adverse Events (participants affected / at risk) | 13/13 | 46/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 (N=13) | Phase 2 (N=50)
Anemia (Blood and lymphatic system disorders) | 0 | 2
Aortic valve disease (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Anal fistula (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Colonic obstruction (Gastrointestinal disorders) | 1 | 0
Colonic perforation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Death NOS (General disorders) | 3 | 4
Fever (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Confusion (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Thromboembolic event (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 (N=13) | Phase 2 (N=50)
Chest pain - cardiac (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Anal pain (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 2 | 1
Bloating (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 4 | 7
Diarrhea (Gastrointestinal disorders) | 1 | 5
Dyspepsia (Gastrointestinal disorders) | 1 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 1
Esophagitis (Gastrointestinal disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 2
Mucositis oral (Gastrointestinal disorders) | 4 | 8
Nausea (Gastrointestinal disorders) | 3 | 2
Rectal pain (Gastrointestinal disorders) | 0 | 2
Rectal ulcer (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Fatigue (General disorders) | 6 | 11
Fever (General disorders) | 0 | 1
Flu like symptoms (General disorders) | 0 | 1
Pain (General disorders) | 2 | 5
Anorectal infection (Infections and infestations) | 0 | 1
Rhinitis infective (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 2
Skin infection (Infections and infestations) | 0 | 2
Upper respiratory infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 3
Alanine aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 5
Lymphocyte count decreased (Investigations) | 0 | 2
Neutrophil count decreased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 1 | 3
Urine output decreased (Investigations) | 0 | 1
Weight loss (Investigations) | 4 | 7
White blood cell decreased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 5 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4
Cognitive disturbance (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 2
Seizure (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 3
Hematuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 9
Urinary retention (Renal and urinary disorders) | 0 | 1
Urinary urgency (Renal and urinary disorders) | 1 | 0
Gynecomastia (Reproductive system and breast disorders) | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 | 20
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 | 1
Hypertension (Vascular disorders) | 3 | 20
Thromboembolic event (Vascular disorders) | 0 | 2
Vascular disorders - Other, specify (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes